CLINICAL TRIAL: NCT06091657
Title: Comparison of Ketamine Plus Dexamethasone Versus Ketamine Alone for Prevention of Severe Shivering After Spinal Anesthesia in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amany Ahmed Eissa, lecturer of anesthesia& ICU, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MS-525-2023
Record Dates: First submitted 2023-10-16; First posted 2023-10-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Intraoperative Shivering; Ketamine With Shivering; Dexamethasone for Shivering; Severe Shivering
Keywords: shivering; ketamine; dexamethasone
MeSH Terms: interventions — Ketamine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine group (Active Comparator): Group K (ketamine):
  syringe (1): the ketamine syringe, dilute 25 mg ketamine in 10 ml saline to have a concentration of 2.5mg/ml. The dose will be 0.25 mg/kg, so we will give 0.1ml/kg of the syringe.
  syringe (2): saline syringe 10 ml saline in 10 ml syringe. (for double blinded technique). we will give 0.1ml/kg of the syringe.
  Interventions: Drug: Ketamine Hydrochloride
- ketamine dexamethasone group (Active Comparator): Group KD (ketamine plus dexamethasone):
  Syringes (1): the ketamine syringe, dilute 25 mg ketamine in 10 ml saline to have a concentration of 2.5mg/ml. The dose will be 0.25 mg/kg, so we will give 0.1ml/kg of the syringe.
  Syringe (2): dexamethasone syringe, 10 mg dexamethasone will be diluted with 10 ml saline in 10 ml syringe, concentration will be 1mg/ml. the dose will be 0.1 mg/kg, so we will give 0.1ml/kg of the syringe.
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — intravenous injection
  Other Names: dexamethasone

SUMMARY:
Shivering is one of the most distressing events of the birth experience for patients. Shivering that occurs with spinal anesthesia is a frequent event, with a reported incidence of up to 50-65%. (1) This may be normal thermoregulatory shivering in response to core hypothermia or may result from the release of cytokines by the surgical procedure. (2-4) shivering is graded with a scale described by Bedside Shivering Assessment Score (BSAS). (3, 4) Most of the literature recommends a variety of non-pharmacological and pharmacological options for the prevention and treatment of shivering after spinal anesthesia. Pethidine, tramadol, clonidine, dexmedetomidine, biogenic amines (serotonin 5-HT3 receptor antagonist), low-dose ketamine, dexamethasone, and magnesium sulfate were used as pharmacological agents. (5) Intravenous (IV) ketamine 0.25 mg/kg was approved as effective in the prevention and treatment of shivering after regional anesthesia and can be used in patients undergoing cesarean sections without adverse effects on the baby. (5) Ketamine is a competitive N-methyl-D-aspartate receptor antagonist, and it is believed that its anti-shivering action is due to non-shivering thermogenesis, either by effect on the hypothalamus or by the β-adrenergic effect of norepinephrine. (6) In spite of the approved effectiveness of ketamine in this issue, moderate to severe shivering (grade ≥ 2) still occurs with an incidence that cannot be ignored. (7-9) Dexamethasone was also approved as an alternative pharmacological agent for the prevention and treatment of mild and moderate shivering. (10) Dexamethasone prevents shivering by regulating immune response and decreasing the temperature gradient between skin and body core via its anti-inflammatory action and inhibition of the release of vasoconstrictors and pyrogenic cytokines. We hypothesize that addition of dexamethasone (0.1 mg\kg) to low dose ketamine (0.25 mg\kg) will be more effective in prevention of severe shivering after spinal anesthesia with cesarean section with minimal sedation of the mother and negligible effect on the baby. This can be applicable in resource-limited settings.

DETAILED DESCRIPTION:
* Preoperatively, a trained anesthetist will assess the patients regarding the age, height; weight. Medical history, medications, laboratory investigation, as well as the patient's airway. Fasting hours will be reviewed(8 hours) In the operating room; temperature will be maintained at 24 °c -26° c by adjusting the temperature setting of the air conditioner.
* Routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied & axillary temperature will be recorded; then intravenous access (18-G cannula) will be inserted and pre-medication ranitidine 40 mg will be administered.
* Baseline vitalsigns will be recorded in the supine position. Ringer lactate infusion (which is kept at room temperature 24°c -26°c) will be started at a rate of 10 ml/kg for the first 30 minutes then reduced to 6 ml/kg till the end of the surgery.

B. drug preparation:

An independent research assistant will be responsible for opening the envelopes and preparing the study drug with no further involvement in the study. The attending anesthetist and data collector will be blinded to the study group.

Group K (ketamine):

syringe (1): the ketamine syringe, dilute 25 mg ketamine in 10 ml saline to have a concentration of 2.5mg/ml. The dose will be 0.25 mg/kg, so we will give 0.1ml/kg of the syringe.

syringe (2): saline syringe 10 ml saline in 10 ml syringe. (for double blinded technique). we will give 0.1ml/kg of the syringe.

Group KD (ketamine plus dexamethasone):

Syringes (1): the ketamine syringe, dilute 25 mg ketamine in 10 ml saline to have a concentration of 2.5mg/ml. The dose will be 0.25 mg/kg, so we will give 0.1ml/kg of the syringe.

Syringe (2): dexamethasone syringe, 10 mg dexamethasone will be diluted with 10 ml saline in 10 ml syringe, concentration will be 1mg/ml. the dose will be 0.1 mg/kg, so we will give 0.1ml/kg of the syringe.

The drugs will be given to the patient by direct intravenous injection through the cannula and flushing with normal saline after administration of the drugs.

Recording of vital signs (arterial blood pressure, heart rate, oxygen saturation axillary temperature) then shifting the patient to the sitting position with a nurse in front of her for administration of subarachnoid block In the sitting posture, a 25G Quincke's spinal needle is used to puncture the L3-L4 interspace under sterile conditions and via the midline route.

After the CSF free flow, 12-15 mg hyperbaric bupivacaine will be givenIntrathecal (according to the patient's height) and the patient will be placed in a supine posture with 15 degrees tilt to left side with a wedge under right iliac bone. Patients will be given 3 liters of oxygen per minute through the nasal cannula.

After spinal anesthesia , arterial blood pressure, heart rate and oxygen saturation will all be recorded immediately after shifting the patient to supine position.

Hypotension is defined as a drop in mean arterial blood pressure (more than 20% below baseline) following spinal injection, and it is treated by increasing intravenous fluid administration and administering 2.5-5 milligrams increments of ephedrine I.V. (every 3-5 minutes) until the hypotension is resolved.

After the sensory block at the level of T4-T6 is confirmed by the lack of sensitivity to cold, surgery will begin. The heart rate, oxygen saturation,are continuously monitored and the blood pressure readings will be taken every 10 minutes till the end of the surgery.

During surgery, a shivering score will be recorded at 15 min intervals and axillary temperature will be recorded after 30 minutes then at the end of the surgery.

Rescue dose of pethidine (25 mg) could be given intravenously if the participant developed grade 3 or grade 4 shivering

* Apgar score of the baby will be recorded as a secondary outcome.
* The level of sedation of the mother using The University of Michigan Sedation Scale (UMSS) will be recorded.

Post operative monitoring:

The participants will be monitored post-operatively for 60 minutes regarding their hemodynamics and shivering score.

Any complications in the Intra operative and post-operative period will be recorded.

1. Measurement tools

* Demographic data as age, sex, BMI, medications, drug allergy and any other comorbidity.
* Heart rate, SpO2, and non-invasive arterial blood pressure will be monitored and recorded before spinal anesthesia and every 10 minutes after spinal anesthesia till the end of the procedure.
* Length of operation and the number of shivering episodes scored ≥2 will be recorded.
* Temperature: axillary temperature will be measured before, immediately and 30 minutes after induction of spinal anesthesia, and at the end of surgery.
* Hemodynamics, temperature, shivering episodes will be recorded for 60 minutes postoperatively.
* Bedside Shivering Assessment Scale shivering score will be recorded at 15 min intervals till the end of the procedure and for 60 minutes in post anesthesia care unit
* Grade 0 if there is no shivering
* Grade 1 if there is no muscle contraction but mild fasciculation of face or neck or peripheral vasoconstriction but no visible shivering
* Grade 2 if there is a visible muscular activity in only one muscle group
* Grade 3 if the muscular activity is in more than one muscle group but not generalized
* Grade 4 if gross muscular activity involving the entire body.
* The level of sedation of the mother will be recorded using The University of Michigan Sedation Scale (UMSS).

Table 1: The University of Michigan Sedation Scale (UMSS)(Liu et al., 2018) Value Patient state 0 • Awake and alert.

1. • Minimally sedated: tired/ sleepy, appropriate response to verbal conversation, and/or sound.
2. • Moderately sedated: somnolent/ sleeping, easily aroused with light tactile stimulation or a simple verbal command.
3. • Deeply sedated: deep sleep, roused only with significant physical stimulation.
4. • Unarousable.

   * .Table 2: Apgar score (Simon et al., 2017) Score 0 points 1 point 2 points Appearance (Skin color) Cyanotic / pale all over Peripheral cyanosis only. Pink Pulse (Heart rate) 0 <100 100-140 Grimace (Reflex irritability) No response to stimulation Grimace or weak cry when stimulated Cry when stimulated Activity (Tone) Floppy Some flexions Well flexed and resisting extension Respiration Apneic Slow, irregular Strong cry

VI. Study outcomes:

1. Primary outcome:

   a) the incidence of shivering attacks intraoperative. ( using Bedside Shivering Assessment Scale)
2. Secondary outcomes:

   1. Apgar score at 1 and 5 minutes, Apgar is a quick test performed on a baby at 1 and 5 minutes after birth. The 1-minute score determines how well the baby tolerated the birthing process. The 5-minute score tells the health care provider how well the baby is doing outside the mother's womb. It also helps measure how well the baby responds if resuscitation is needed right after birth.
   2. Intraoperative hemodynamics assessment Immediately after injection of the medications and every 10 minutes till the end of the procedure including: heart rate, arterial blood pressure and number of hypotensive episodes
   3. Sedation of the mother immediately after injection of drug and after 30 minutes using The University of Michigan Sedation Scale (UMSS)

ELIGIBILITY:
Inclusion Criteria:

* 1. Inclusion criteria

  * pregnant females
  * aged 18 to 45 years
  * ASA physical status II
  * elective Cesarean sections under spinal anesthesia

    2. Exclusion criteria
  * Contraindications for spinal anesthesia
  * Emergency cesarean sections
  * Patient with initial body temperature >38°c or <36°c
  * Allergy to any of the drugs used in the study
  * Pre Existing neurological diseases (particularly those that wax and wane, e.g.multiple sclerosis)
  * Thrombocytopenia and coagulation disorders.
  * Severe stenotic heart disease.

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
number of shivering episodes | the whole procedure and for 60 minutes postoperative
  ● the number of shivering episodes scored ≥3 will be recorded.

SECONDARY OUTCOMES:
sedation score of the mother | 120 minutes
APGAR score of the baby | 5 minutes
hemodynamics | 120 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Aini Hospitals, Cairo, Egypt